CLINICAL TRIAL: NCT06122610
Title: Dosimetry-Guided 177Lu-DOTATATE Treatment Planning Using 64Cu-DOTATATE as a Surrogate
Brief Title: Using Novel Imaging to More Safely Treat Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0121; Protocol Version 12/12/2025 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison)
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Tumors; Somatostatin Receptor-positive Neuroendocrine Tumor
Keywords: neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Tomography, Emission-Computed, Single-Photon; Tomography, X-Ray Computed; Single Photon Emission Computed Tomography Computed Tomography; Positron Emission Tomography Computed Tomography; 64Cu-DOTATATE; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Participants treated with Lutathera (Experimental)
  Interventions: Device: Single Photon Emission Computed Tomography/ Computed Tomography (SPECT/CT); Device: Photon Emission Tomography / CT (PET/CT); Drug: 64Cu-Dotatate; Drug: 177Lu-Dotatate

INTERVENTIONS:
Device: Single Photon Emission Computed Tomography/ Computed Tomography (SPECT/CT) — SPECT/CT will be performed after first cycle of Lutathera® treatment
Device: Photon Emission Tomography / CT (PET/CT) — PET/CT will be performed after 64Cu-DOTATATE and Lutathera® treatment
Drug: 64Cu-Dotatate — Standard of care administration of radioactive drug for PET/CT
  Other Names: Detectnet
Drug: 177Lu-Dotatate — Standard of care administration of radioactive drug for PET/CT and SPECT/CT
  Other Names: Lutathera®

SUMMARY:
The goal of this research is to determine if DetectnetTM PET/CT can be used to make Lutathera therapy safer for patients with neuroendocrine cancer.

Participants will:

* Complete two phases involving 6 visits
* Undergo additional research PET/CT, and possibly SPECT/CT scans

DETAILED DESCRIPTION:
The goal of this research study is to determine if DetectnetTM PET/CT scanning over several days can be used to deliver Lutathera in a safer manner.

In this research, participants will be asked to complete a screening phase and possibly a dosimetry phase. The screening phase will require 2 visits. The dosimetry phase will also require 3 research visits.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for 177Lu-DOTATATE (Lutathera) treatment for somatostatin receptor-positive neuroendocrine tumor

Exclusion Criteria:

* Unable to lie flat during or tolerate PET/CT or SPECT/CT
* Known incompatibility to CT. SPECT, or PET scans
* Unlikely to comply with study procedures, restrictions and requirements and judged by the investigator that the participant is not suitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Compare pre-therapy and post-therapy voxel-based dosimetry estimates | Baseline and 120 hours post-dose
  Absorbed doses to organs will be estimated using radiation dosimetry methods based on both multi-timepoint PET and multi-timepoint SPECT imaging. Mean dose estimates in units of Gy to the index tumor(s) and dose limiting organs (kidneys and bone marrow) will be compared between PET-based dosimetry and SPECT-based dosimetry. Using SPECT-based dosimetry as the gold standard truth, Bland-Altman analysis will be performed for each organ/tumor to compare PET-based dose estimates to SPECT-based estimates. Mean bias and 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Absorbed radiation doses | 1 hour post-dose, 4 hours post-dose, 48 hours post-dose, 120 hours post-dose
  Absorbed radiation doses from 177Lu-DOTATATE in organs will be summarized with descriptive statistics.
Absorbed radiation doses of 64Cu-DOTATATE | 1 hour post-dose, 4 hours post-dose, 48 hours post-dose, 120 hours post-dose
  Absorbed radiation doses of 177Lu-DOTATATE in organs using 64Cu-DOTATATE as an imagining surrogate will be summarized with descriptive statistics.
Compare 3D voxel-based versus model based dosimetry in participants receiving 177Lu_DOTATATE | Baseline and 120 hours post-dose
  Absorbed doses to organs will be estimated using radiation dosimetry methods based on multi-timepoint SPECT imaging. Mean dose estimates in units of Gy to the index tumor(s) and dose limiting organs (kidneys and bone marrow) will be compared between 3D voxel-based and model-based dosimetry methods. Using 3D voxel-based dosimetry as the gold standard truth, Bland-Altman analysis will be performed for each organ/tumor to compare 3D voxel-based to model-based methods. Mean bias and 95% confidence intervals will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Changhee Lee, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No